CLINICAL TRIAL: NCT03523832
Title: Preemptive Analgesia in Total Knee Arthroplasty: Comparing the Effects of Single Dose Combined Celecoxib With Pregabaline and Repetition Dose Combined Celecoxib With Pregabaline (Double Blind Controlled Clinical Trial)
Brief Title: Preemptive Analgesia in Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 04
Record Dates: First submitted 2018-04-17; First posted 2018-05-14 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2018-04

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): celecoxib 400mg and pregabaline 150mg 1 hour before operation
  Interventions: Drug: Celecoxib and Pregabaline
- Group 2 (Active Comparator): celecoxib 200mg and pregabaline 75mg twice daily started from 3 days before operation
  Interventions: Drug: Celecoxib and Pregabaline
- Group 3 (Placebo Comparator): No treatment given
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Celecoxib and Pregabaline — Single dose versus repetition dose
  Arms: Group 1; Group 2
Other: Placebo — Placebo
  Arms: Group 3

SUMMARY:
Acute Pain is the most common early complication after total knee arthroplasty that caused delayed mobilization, demands of morphine, and higher operative cost. There were many researches that had been done in analgesia method to find the most effective analgesia, lowest side effect, and easy to apply. Preemptive analgesia of combined celecoxib and pregabalin were reported to give a promising outcome.

In a randomized, double blind controlled clinical trial, 30 subjects underwent surgery for total knee arthroplasty using 15-20mg bupivacaine 5% epidural anesthesia. All subjects were divided into three groups. First group was given celecoxib 400mg and pregabaline 150mg 1 hour before operation, second group was given celecoxib 200mg and pregabaline 75mg twice daily started from 3 days before operation, and the last group was given placebo. The outcome was measured with VAS, knee ROM, and post-operative mobilization

ELIGIBILITY:
Inclusion Criteria:

* 55-80 years old patients who come to orthopaedic polyclinic
* underwent TKA procedure
* have osteoarthritis
* consumed pain killer and anti inflamatory drugs routinely

Exclusion Criteria:

* psychiatric disorder
* have history of renal disease
* histroy of chronic neurophatic
* have genu arthritis that caused by rheumatid arthritis and infection
* diabetic and obesity
* coagulopathy
* patients with severe pain that needed immediate analgesia regimen

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Total Morphine Consumption | Third day post-operative
  In this study, morphine is given by patient control analgesia (PCA).

SECONDARY OUTCOMES:
Post-operative Pain | every morning [daily], up to 3 days
  Measured and evaluated by Visual Analogue Scale (VAS). VAS score of 1-10. With the maximal of 10. Ranging from no pain to unbearable pain. Worst pain is in score 10.
Knee functional outcome | every morning [daily], up to 3 days
  Measured by active knee range of motion using goniometer. The outcome scale is in degree range of motion. The knee range of motion is 0 degree (total extension) to 135 degree (full flexion). The more range of motion degree, the better the result.
Mobilization | on the first day, standing on the second day, and walking on the third day
  The patient is expected to be able to do sitting motion

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lubis AMT, Rawung RBV, Tantri AR. Preemptive Analgesia in Total Knee Arthroplasty: Comparing the Effects of Single Dose Combining Celecoxib with Pregabalin and Repetition Dose Combining Celecoxib with Pregabalin: Double-Blind Controlled Clinical Trial. Pain Res Treat. 2018 Aug 7;2018:3807217. doi: 10.1155/2018/3807217. eCollection 2018. PMID 30174951

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT03523832/Prot_SAP_000.pdf